CLINICAL TRIAL: NCT04932603
Title: Impact of Multidisciplinary Team Approach on the Utilization and Risks Related to Antithrombotic Drugs in Older Patients With Atrial Fibrillation
Brief Title: Multidisciplinary Team Approach to Prescribe Antithrombotic Therapy in Older People With Atrial Fibrillation
Acronym: ANTITHROMBOTEA
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP210392
Record Dates: First submitted 2021-06-14; First posted 2021-06-21 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-07

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Frail Elderly; Anticoagulants; Platelet Aggregation Inhibitors; Multidisciplinary team
MeSH Terms: conditions — Atrial Fibrillation | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- experimental: Patients with AF, hospitalized in one of the 6 geriatrics units participating in the study, aged 75 years or over, without evaluation of their antithrombotic treatment by the multidisciplinary team. The lack of review of patient's file by the multidisciplinary team is based on physician decision.
  Interventions: Other: Standard of care, with intervention of the multidisciplinary team
- Standard of care

INTERVENTIONS:
Other: Standard of care, with intervention of the multidisciplinary team — Patients with AF, aged of 75 years or more, with evaluation of their antithrombotic treatment by the multidisciplinary team. The review of patient's file by the multidisciplinary team is based on physician decision. These patients are hospitalized in one of the 6 geriatrics units participating in the study and / or are hospitalized in another ward but their clinical file is reviewed by the multidisciplinary team.
  Groups: experimental

SUMMARY:
Antithrombotic drugs, which include antiplatelet and anticoagulant therapies, are used to prevent and treat many cardiovascular disorders. With the increase in prevalence of cardiovascular diseases and medical progress, these treatments are increasingly being prescribed, particularly in older patients. One of the main indications of antithrombotic drugs is atrial fibrillation (AF), a disease highly prevalent in older people, a population at high risk of adverse drug events. Notably, antithrombotic drugs are the first involved in serious adverse drug events, among which 40-70% may be preventable. In this context, six units of the hospital group "Assistance Publique - Hôpitaux de Paris" have created a multidisciplinary team which assesses antithrombotic prescriptions in older patients with AF. This team, gathering geriatricians, cardiologists, neurologists and haematologist specialized in haemostasis, evaluates the patient medical profile and suggests the most appropriate antithrombotic treatment based on their expertise and the available recommendations. Here we want to look at patients outcomes in light of the intervention of this multidisciplinary team.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the impact of the multidisciplinary team on the composite outcome of all-cause mortality, ischemic event or bleeding event at 3 months. Secondary objectives are to evaluate this composite outcome at 6 months and all-cause mortality, occurrence of ischemic event, occurrence of bleeding event, at 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* 75 years old patients or more
* Diagnosis of AF
* Hospitalized in one of the 6 geriatrics unit participating in the study and / or whose clinical file is reviewed by the multidisciplinary team

Exclusion Criteria:

* opposition to data collection for research purposes

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients hospitalized in 6 geriatrics units in the Greater Paris area and / or whose clinical file is reviewed by the multidisciplinary team PAtiet
Sampling Method: Non-Probability Sample
Enrollment: 833 (Actual)
Dates: Start 2021-05-29 (Actual); Primary Completion 2024-07-05 (Actual); Study Completion 2024-07-05 (Actual)

PRIMARY OUTCOMES:
Composite outcome of all-cause mortality, ischemic event or bleeding event | 3 months after inclusion
  All-cause mortality will be assess using patient's medical record or reported death by the referent general practitioner. Ischemic events include acute coronary syndrome, transient ischemic stroke or permanent ischemic stroke, arterial embolism, deep vein thrombosis and pulmonary embolism. Bleeding events include any bleeding event requiring a medical consult or a hospitalization

SECONDARY OUTCOMES:
All-cause mortality | 3 months after inclusion
  All-cause mortality will be assess using patient's medical record or reported death by the referent general practitioner.
Ischemic event | 3 months after inclusion
  Ischemic events include acute coronary syndrome, transient ischemic stroke or permanent ischemic stroke, arterial embolism, deep vein thrombosis
Ischemic event | 6 months after inclusion
  Ischemic events include acute coronary syndrome, transient ischemic stroke or permanent ischemic stroke, arterial embolism, deep vein thrombosis
Bleeding event | 3 months after inclusion
  Bleeding events include any bleeding event requiring a medical consult or a hospitalization.
Bleeding event | 6 months after inclusion
  Bleeding events include any bleeding event requiring a medical consult or a hospitalization.
Composite outcome of all-cause mortality, ischemic event or bleeding event | 6 months after inclusion
  All-cause mortality will be assess by patient's medical record or reported death by the referent general practitioner. Ischemic events include transient ischemic attack or ischemic stroke, arterial embolism, deep vein thrombosis and pulmonary embolism. Bleeding events include any bleeding event requiring a medical consult or a hospitalization.
All-cause mortality | 6 months after inclusion
  All-cause mortality will be assess by patient's medical record or reported death by the referent general practitioner.

CONTACTS AND LOCATIONS:
Locations (1):
- Unité de gériatrie aiguë, hôpital Pitié-Salpêtrière (Pr Marc Verny), Paris, France

REFERENCES:
- [Derived] Prunel M, Cochard A, Abbas L, Baudry E, Pautas E, Legris N, Assayag P, Frere C, Verny M, Simon-Tillaux N, Zerah L. Multidisciplinary team for antithrombotics management and clinical outcomes in older adults with atrial fibrillation: a target trial emulation. BMC Med. 2025 Sep 29;23(1):521. doi: 10.1186/s12916-025-04291-9. PMID 41024059